CLINICAL TRIAL: NCT05192551
Title: Comparison of Patient Satisfaction and Efficacy of Different PEG-based Bowel Preparations- an Observational Study in Five Endoscopy Units in Sweden
Brief Title: Patient Satisfaction and Efficacy of Different PEG-based Bowel Preparations- an Observational Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Perjohan Lindfors, MD, PhD, Karolinska Institutet
Other Study IDs: Bowelprep
Record Dates: First submitted 2021-12-07; First posted 2022-01-14 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Patient Satisfaction and Efficacy of Bowel-preparation
Keywords: Bowel-prep; Colonoscopy; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Polyethylene Glycols

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Plenvu: A new type of low-volume bowel-prep recently approved and introduced in the Swedish market. The dose is 500 ml x 2, The first dose is given the evening before the colonoscopy and the second dose is given 4-5 hours before the colonoscopy.
  Interventions: Other: Bowel-prep (Plenvu as experimental arm)
- Laxabon: A standard high volume bowel-prep, used for a long time in Sweden. The dose is 2000 ml x 2. The first dose is given the evening before the colonoscopy and the second dose is given 4-5 hours before the colonoscopy.
  Interventions: Other: Bowel-prep (Plenvu as experimental arm)
- Vistaprep: A standard high volume bowel-prep, used for a long time in Sweden. The dose is 2000 ml x 2. The first dose is given the evening before the colonoscopy and the second dose is given 4-5 hours before the colonoscopy.
  Interventions: Other: Bowel-prep (Plenvu as experimental arm)
- Movprep: A standard median volume bowel-prep, used for a long time in Sweden. The dose is 1000 ml x 2. The first dose is given the evening before the colonoscopy and the second dose is given 4-5 hours before the colonoscopy.
  Interventions: Other: Bowel-prep (Plenvu as experimental arm)

INTERVENTIONS:
Other: Bowel-prep (Plenvu as experimental arm) — In this study we will investigate the efficacy and patient satisfaction of the,in Sweden recently approved and introduced low-dose, Peg-based bowel-prep Plenvu in comparsion with the standard bowel-preps used i today's clinical routine
  Other Names: Laxabon,; Vistaprep; Movprep

SUMMARY:
An multi-center, observational study where we compare the current standard, PEG-based bowel-prep to a (in Sweden) recently approved and introduced low volume (1 litre) PEG-based bowel-prep (Plenvu) in a clinical routine situation.

The investigators will investigate if there are any differences in patient satisfaction and efficacy of the different bowel preparations

DETAILED DESCRIPTION:
When performing Colonoscopy it is essential to use a bowel-prep that is highly effective and at the same time tolerable to intake for the patient to ensure that the patients intakes the recommended amount of the bowel-prep.

This in order to be able to detect pathological findings in the mucosa. Currently in n Sweden the standard bowel-prep used in most endoscopy-units is high volume bowel preps (4 litres) in split dose. It can be difficult for the patient to intake the whole dose wish can lead to a sub-optimal bowel-cleansing.

Recently, in Sweden, a new low-volume bowel-prep has been approved and introduced (Plenvu).

This preparation, totally 1 litre of bowel prep given in a split dose is potentially easier for the patient to intake but it is essentially to ensure that the efficacy i at least as good as the current high dose preparation. In this study the investigators will therefore investigate patient satisfaction and efficacy of the different bowel preparations, comparing Plenvu with the current standard bowel-prep regime at the participating endoscopy units.

Five endoscopy units participates in this study (Endoskopi City, Stockholm, Endoskopienheten i Malmö, Endoskopienheten i Linköping, Endoskopienheten i Örebro, Endoskopienheten Ersta sjukhus, Stockholm).

In each endoscopy unit 100 consecutive patients will be prescribed Plenvu and another 100 consecutive patients will be prescribed the current standard bowel-prep at the actual unit. a total of 1000 patients will participate in the study.

The currently used bowel-preps at the different endoscopy units are: Vistaprep, Laxabon and Movprep This is a study performed in a clinical context and no randomization is made. When arriving to the endoscopy unit patients are asked to participate in the study and if willing to participate patients will sign an informed consent-form.

Before the colonoscopy the patients fills in a questionnaire about the bowel-prep experience concerning; smell, taste, overall experience (five graded scales) of the prep. In the questionnaire patients are also asked how much of the prescribed bowel-prep that have been digested and how much extra fluid the patient have been drinking during the preparation process. The patients are also asked about if they have been experienced nausea or been vomiting.

After the colonoscopy, the gastroenterologist performing the endoscopy fills in the Boston Bowel Preparation Scale (BBPS) as a measure of how successful the bowel cleansing has been.

Based on this information the investigators will compare patient satisfaction and efficacy of the bowel-cleansing in the group that has been prescribed Plenvu to the group that has been prescribed the endoscopy-units standard bowel-prep

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 admitted for colonoscopy at the participating endoscopy-units.

Exclusion Criteria:

* Renal failure or other contraindication for using low-dose bowel-preps
* not speking or reading swedish
* Need for a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled for a routine colonoscopy at the endoscopy unit
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with bowel prep | Day 1,When arriving to the endoscopy unit, Immediately before the endoscopy
  When arriving to the endoscopy unit the patients fills in a questionnaire about their bowel-prep experience concerning; smell, taste, overall experience (five graded scales) of the prep. The higher the number are the more satisfied the patient are with the current experience (smell, taste and overall experience.
  In the questionnaire they are also asked how much of the prescribed bowel-prep they have digested and how much extra fluid they have been drinking during the preparation process (0-4 litres).
Efficacy of the bowel prep | Day 1,Directly after the colonoscopy,
  Immediately after the colonoscopy the gastroenterologist who has performed the investigation fills in the Boston Bowel Preparation Scale,a widely used scale describing how clean the bowel is in each of the three segment ant in total. Each segment is graded form 0-3 (3 perfect cleaning) and a sum-score of 0-9 (9 perfect clening) is calculated. The higher the number the better the cleansing are

SECONDARY OUTCOMES:
Differences in the reported frequency of nausea and vomiting during the bowel-preparation process | Day 1,When arriving to the endoscopy unit, Immediately before the endoscopy
  The patients are asked if they have been experienced nausea or been vomiting (yes /no)

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Universitetssjukhuset Linköping, Linköping
  - Skåne Universitetssjukhus, Malmo
  - Universitetssjukhuset Örebro, Örebro
  - Aleris GastromottagningenCity, Stockholm
  - Ersta sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: No